CLINICAL TRIAL: NCT06030388
Title: STrength and AeRobic Training Against Vasomotor Symptoms (START) in Postmenopausal Women
Brief Title: Strength and Aerobic Training Against Hot Flushes in Postmenopausal Women
Acronym: START
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Region Östergötland (Other); Länssjukhuset i Kalmar län (Other Government)
Responsible Party: Principal Investigator, Anna-Clara Spetz Holm, Associate professor, Medical Doctor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: START2022-05030-1
Record Dates: First submitted 2023-06-15; First posted 2023-09-11 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Postmenopausal Symptoms; Hot Flashes
Keywords: aerobic training; strength training
MeSH Terms: conditions — Hot Flashes | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Three-armed randomised trial where participants are randomised to 1) strength training, 2) high-intensity aerobic training or 3) untreated control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Strength training (Active Comparator): Standardised programme with the following exercises: chest press, leg press, row, leg curl, latissimus dorsi pull down and leg extension in seated resistance machines. Training will be preceded by 7-10 minutes of warm-up and followed by two body-weight exercises for the abdominal and back muscles for two sets as many repetitions as possible, and thereafter cool down and stretches. The set-up of each machine will be recorded in the training diary.
  Weeks 1-3 will include two sets of training with 15-20 repetition-maximum (RM) and weeks 4-15 two sets with 8-12 RM. Throughout the intervention, loads will be adjusted to achieve muscle fatigue and approach training to failure during each set with the intent to maximize beta-endorphin release.
  Interventions: Other: Strength training
- High-intensity aerobic training (Active Comparator): Participants will be recommended to attend spinning classes three times per week. During their first visit to the training venue, they will meet a sports physiotherapist or personal trainer to be introduced to the spinning bike intervention. The intended intensity is ≥ 14 on the Borg rating of perceived exertion scale, equivalent to high intensity training (>70% of VO2max) with the aim of attaining sufficient stimulus for beta-endorphin release. During weeks 1-3 participants will attend spinning classes for beginners with lower intensity and predominantly seated cycling. They will progress to higher intensity classes with greater variation between seated and standing cycling during week 4-15.
  Interventions: Other: High-intensity aerobic training
- Control group (No Intervention): The control group will be recommended to carry on physical activity as usual and not to change their training or dietary habits during the 15-week study period. The control group will be contacted every fourth weeks by a research nurse to follow up on their general well-being and any questions they might have about menopause. After the study period they will be offered individual advise about training from a physiotherapist or personal trainer.

INTERVENTIONS:
Other: Strength training — Both interventions (strength training and high intensity aerobic training) will be introduced with a 3-week adaptation period with lower loads (strength training) or intensity (aerobic training) followed by a 12-week period on the intended load/intensity. All participants in the intervention groups will be recommended to exercise three times per week (one hour per session) and in addition be active with everyday low-intensity physical activity. A structured and detailed training diary will be used in both groups to register frequency of each training session, as well as everyday physical activity. For the strength training, load and dose will also be registered for each training session.
  Arms: Strength training
Other: High-intensity aerobic training — Both interventions (strength training and high intensity aerobic training) will be introduced with a 3-week adaptation period with lower loads (strength training) or intensity (aerobic training) followed by a 12-week period on the intended load/intensity. All participants in the intervention groups will be recommended to exercise three times per week (one hour per session) and in addition be active with everyday low-intensity physical activity. A structured and detailed training diary will be used in both groups to register frequency of each training session, as well as everyday physical activity. For the strength training, load and dose will also be registered for each training session.
  Arms: High-intensity aerobic training

SUMMARY:
The goal of this randomised controlled trial is to investigate the effects of and compare two modes of physical exercise (strength training and high-intensity aerobic exercise) to unchanged physical activity on vasomotor symptoms (hot flushes) in postmenopausal women. The main question it aims to answer is the effect of 15 weeks of strength training vs high intensity aerobic training vs unchanged physical activity on frequency and severity of hot flushes. Participants will be randomised to:

1. strength training
2. high-intensity aerobic training
3. untreated control group.

Researchers will compare strength training, high-intensity aerobic training and untreated control group to see if training can reduce hot flushes.

DETAILED DESCRIPTION:
The overall aim is to investigate the efficacy of and compare two modes of physical exercise (strength training and high-intensity aerobic exercise) to unchanged physical activity on vasomotor symptoms (VMS), as well as secondary outcomes such as health-related quality of life, sleep quality, physical activity levels, clinical outcomes, biomarkers, bone markers (outcome added January 2025), bone mineral density (outcome added January 2025), perceptions of and adherence to the interventions. In a longer perspective, the goal is to find evidence-based treatment options for VMS in postmenopausal women that are safe and effective, and have positive effects on health and quality of life after menopause.

Our hypothesis is that strength training and high-intensity aerobic exercise will reduce VMS in postmenopausal women and improve quality of life as well as clinical outcomes more than in a control group with unchanged physical activity. We also hypothesize that strength training and high-intensity aerobic training will have the same effect on the primary outcome (change in VMS) and that most of the changes in secondary outcomes will be superior in the high-intensity aerobic training group compared to the strength training group.

This is an open, two-centre, parallel, randomized controlled study performed according to the SPIRIT and CONSORT statements

Recruitment will take place by advertising on social media, in local newspapers and in the Women's clinics and primary care centers in Linköping and Kalmar. Women who respond to the advertisements will be contacted by a member of the research group or research nurse to receive information about the study and screen for inclusion and exclusion criteria. Women who are possibly eligible will be invited to a screening visit for further information and informed consent. At the visit, inclusion and exclusion criteria will be checked by a physician, and a clinical examination will be performed. Eligible participants will receive a VMS screening diary and invited to a second visit 2-3 weeks later where inclusion and randomization will be performed if the VMS inclusion criteria are fulfilled.

Randomization An allocation sequence using a computerized random number generator will be prepared by a statistician not involved in recruitment. Opaque sealed and sequentially numbered envelopes with group allocation will be prepared and opened in the presence of the participant upon inclusion and randomization.

Power analysis: A sample size calculation was made based on the results of our previous study on strength training for VMS (Berin et al 2019) and showed that to detect a 50% difference in moderate and severe hot flushes with 80% power and expected dropout rate of 20% 40 participants in total would be needed. For this three-armed set-up we estimate that 20 participants in each group will be needed, i.e. 60 in total. To also achieve sufficient power for some of the secondary outcomes the intended sample size is increased to 30 per group, 90 in total.

Data analysis: The primary analysis will be performed according to the intention-to-treat principle, including all participants who provided more than baseline data for the primary outcome. For quantitative interval data mixed design ANOVAs will be used to analyze the effect over time between and within groups. For the between-group comparisons effect sizes will be calculated. For ordinal data, such as the questionnaires, Kruskal-Wallis and Friedman test will be used for statistical analysis of the effect. Participants who complete two or more training sessions per week will be considered adherent with their assigned intervention and included in a per-protocol analysis. Detailed description of adherence, such as the fidelity with the training interventions, will be presented descriptively.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (one of: ≥ 12 months since last menstruation; amenorrhea due to intrauterine device or hysterectomy and Follicle Stimulating Hormone (FSH) >30 mIU/ml; bilateral oophorectomy; induced menopause due to chemotherapy or radiation and ≥2 years amenorrhea);
* ≥ 28 moderate to severe hot flushes per week during a 2-week screening period, registered through a daily VMS diary;
* Age ≥45 years;
* Physical ability to participate in strength training or high intensity aerobic exercise for 60 minutes, 3 times/week during 15 weeks;
* Understand Swedish orally and in writing

Exclusion Criteria:

* Regular physical activity >30 minutes per week of vigorous intensity or ≥150 minutes of moderate intensity or combined activities representing maximum 150 minutes of moderate intensity;
* Use of systemic menopausal hormone therapy the last 2 months;
* Use of natural preparations such as herbal preparations for VMS, or other medications for VMS the last 2 months;
* Capillary hemoglobin <110 g/l;
* Blood pressure >160 mmHg systolic or >100 mmHg diastolic;
* Unstable medical condition with a potential to affect VMS (like unregulated thyroid disease);
* Medical condition that by a physician is judged not appropriate (because of potential to affect VMS or risk of injury with vigorous exercise)

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of moderate and severe hot flushes | baseline to 15 weeks
  Frequency of hot flushes per 24 h daily recorded in hot flush diary from baseline throughout 15 weeks of intervention.

SECONDARY OUTCOMES:
Frequency of moderate and severe hot flushes | baseline to 6 months, 1, 2 and 5 years
  Frequency of hot flushes per 24 h daily recorded in hot flush diary 2 weeks at baseline and 2 weeks at each of the time points.
Severity of hot flushes | baseline to 15 weeks, 6 months, 1, 2 and 5 years
  Severity of hot flushes per 24 hours recorded in hot flush diary from baseline throughout 15 weeks of intervention and two weeks during follow-up.
Generic health-related quality of life | baseline to 15 weeks, 6 months, 1, 2 and 5 years after intervention
  Short-form 36, 36 questions in 8 scales. Scores for each domain range from 0-100, and a high score represents a higher health-related quality of life.
Women specific health-related quality of life | baseline to 15 weeks, 6 months, 1, 2 and 5 years after intervention
  Women's health questionnaire nine sub-scales with four-point scales (yes definitely, yes sometimes, not not much, no not at all) that are reduced to binary options (0/1). The subscale items are summated and divided by the number of items in each subscale.A higher score represents worse outcome.
Physical activity levels | baseline to 15 weeks, 6 months, 1, 2 and 5 years after intervention
  International Physical Activity Questionnaire short form, the participant describes the amount of time (minutes and hours) that is spent on different physical activities each week, the more time, the better, except for the question about the amount of time spent in sitting.
Sleep quality | baseline to 15 weeks, 6 months, 1, 2 and 5 years after intervention
  Pittsburgh sleep quality index, 7 domains. For the total instrument, the lower score, the better, from 0 (best) to 21 (worst).
Diet | baseline to 15 weeks, 6 months, 1, 2 and 5 years
  Bespoke questionnaire, primarily to control for changes during the intervention period. Registration of amounts or portions. Results are presented question by question descriptively.
Accomplished physical activity | baseline to 15 weeks, 6 months, 1, 2 and 5 years after intervention
  Bespoke training diary
Bioimpedance | baseline to 15 weeks
  Fat mass (%) and fat-free (muscle) mass (%)
Weight | baseline to 15 weeks
  kilogram (kg)
Lenght | baseline to 15 weeks
  meters (m)
Body mass index | baseline to 15 weeks
  kilograms/meters2 (kg/m2)
Waist circumference | baseline to 15 weeks
  millimeters (mm)
Systolic and diastolic blood pressure | baseline to 15 weeks
  Unit millimetre of mercury (mmHg)
Hematologic and ironstatus changes | baseline to 15 weeks, and 1 year
  Hemoglobin full body count, Transferrin(gram/Litre), and Ferritin (microgram/Litre)
Changes in blood-lipids | baseline to 15 weeks, and 1 year
  apolipoprotein A1, apolipoprotein B (gram/Litre) and total cholesterol, low-density lipoprotein, high-density lipoprotein (mmol/L) and leptin (ng/mL)
Changes in sex hormones and gonadotrophins | baseline to 15 weeks, and 1 year
  Estradiol (pmol/Litre), Sex hormone bindning globulin, Testosterone (nmol/Litre), follicle-stimulating hormone, luteinizing hormone (IE/Litre)
Changes in glucose profile | baseline to 15 weeks, and 1 year
  HbA1c (mmol/Litre) and fasting blood glucose (mmol/L)
Changes in inflammatory biomarkers | baseline to 15 weeks, and 1 year
  high-sensitive C-reactive Protein (microgram/Litre), Brain-derived neutrophic factor, Matrix metalloproteinase-2 and -9 (ng/mL), Interleukin -4, -6, -7, -8, 10, -15, tumour necrosis factor, monocyte chemoattractant protein-1 (pg/mL)
Changes in the lenght of telomeres in white blood cells | baseline to 15 weeks, and 1 year
  Telomeres (kilobase) pair
Changes in bone markers | Baseline to 15 weeks, and 1 year
  25-hydroxyvitamin D (25OHD) (nmol/L), Parathyroid hormone (PTH) (pmol/L), C-terminal telopeptide cross-links of collagen type I (CTX) (ng/L), Tartrate-resistant acid phosphatase isoform 5B (TRACP5B) (U/L), Type I procollagen intact N-terminal propeptide (PINP) (µg/L), Bone-specific alkaline phosphatase (BALP) (µg/L or U/L (assay dependent)), Bioactive sclerostin (pmol/L), Osteoprotegerin (OPG) (pmol/L), Free soluble receptor activator of nuclear factor κB ligand (RANKL) (pmol/L), Intact fibroblast growth factor 23 (FGF23) (pg/mL), Irisin (µg/L). Measurement added in January 2025 and data was only collected for participants entering the study from January 2025.
Change in body composition (DXA - dual energy x ray absorptiometry) | Baseline to 15 weeks
  Fat mass, lean mass. Measurement added in January 2025 and data was only collected for participants entering the study from January 2025.
Change in bone mineral density (DXA - dual energy x ray absorptiometry) | Baseline to 15 weeks
  Bone mineral density (g/area) and T-score in spine and hip. Measurement added in January 2025 and data was only collected for participants entering the study from January 2025.
Change in exercise capacity | baseline to 15 weeks
  Change in exercise capacity is primarily used as a measure of adherence and obtained through cardiopulmonary exercise testing assessing maximum oxygen uptake milliliter/kilogram/minute (ml/kg/minute) and analysed according to local clinical routines.
Experiences of the interventions, facilitators and barriers | baseline to 15 weeks
  Bespoke questionnaire, only for intervention groups. Results will be presented descriptively question by question.
Adherence to the interventions | baseline to 15 weeks
  Assessed through bespoke training diary where each training session is registered and the total number of training sessions as well as training sessions/week will be calculated.
Muscle strength | baseline to 15 weeks
  For strength training group only, measured using 8 repetition-maximum tests.
Adverse events | baseline to 15 weeks
  Adverse events of taking part in the study

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Clara Spetz Holm, Ass prof, MD, Principal Investigator — Region Östergötland, Linköping university
Locations (2):
- Sweden (2):
  - Region Kalmar Län, Kalmar
  - Region Östergötland, Linköping

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in publications may be available upon reasonable request to the principal investigator
Time Frame: 1 year after publication.

REFERENCES:
- [Background] Berin E, Hammar M, Lindblom H, Lindh-Astrand L, Ruber M, Spetz Holm AC. Resistance training for hot flushes in postmenopausal women: A randomised controlled trial. Maturitas. 2019 Aug;126:55-60. doi: 10.1016/j.maturitas.2019.05.005. Epub 2019 May 14. PMID 31239119